CLINICAL TRIAL: NCT06606652
Title: Effect of Acute Caffeine Intake on Muscle Electrical Activity and Muscular Strength, Power, and Endurance Performance
Brief Title: Caffeine, Resistance Exercise and EMG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Alberto Pérez-López, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: CEIP/2023/4/093_2
Record Dates: First submitted 2024-09-09; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Caffeine
MeSH Terms: interventions — Caffeine

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Caffeine - Morning (Experimental)
  Interventions: Dietary Supplement: Caffeine
- Caffeine - Evening (Experimental)
  Interventions: Dietary Supplement: Caffeine
- Placebo - Morning (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo
- Placebo - Evening (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Caffeine — Acute caffeine intake (3 mg/kg)
  Arms: Caffeine - Evening; Caffeine - Morning
Dietary Supplement: Placebo — Acute placebo intake (3 mg/kg of maltodextrin)
  Arms: Placebo - Evening; Placebo - Morning

SUMMARY:
Introduction: Several studies have evaluated and confirmed the ergogenic effects of acute caffeine intake on sports performance. However, some studies suggest that this effect predominantly occurs in large muscle groups, potentially due to increased skeletal muscle electrical activity.

Objectives: This study aims to evaluate the acute effects of caffeine intake on strength, power, muscle endurance, and muscle electrical activity in young adults. It will also analyze the influence of circadian rhythms (morning vs. afternoon) on exercise performance (bench press vs. squat).

Methods: Twelve healthy, physically active participants will be recruited for the study. Using a triple-blind, crossover, randomized, and controlled design, participants will ingest either caffeine (3 mg/kg body mass) or a placebo (maltodextrin, 3 mg/kg) 60 minutes before the trial. Muscular strength, power, and endurance performance will then be assessed through 1RM tests, and at 25%, 50%, 75%, and 90% of 1RM, along with muscle endurance tests at 65% of 1RM, for both squat and bench press exercises. EMG will be used to measure skeletal muscle electrical activity during the tests. The experimental sessions will be conducted in the morning (8:00 am to 10:00 am) and the afternoon (4:30 pm to 6:30 pm).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 35 years.
* Body Mass Index (BMI) < 25 kg/m².
* Resistance-trained individuals (more than 2 years of structured training).
* Healthy men and women without neurological, cardiometabolic, immunological, or physical conditions that prevent them from exercising.
* Participants must be able to perform the tests described in the following section.

Exclusion Criteria:

* History of neuromuscular diseases, heart disease, or conditions that may affect liver or muscle metabolism.
* Use of drugs, stimulants, or sports supplements that could interfere with the dietary supplement used in the study.
* Sedentary habits (less than 150 minutes/week of moderate exercise).
* Having undergone prolonged periods of physical inactivity in the 6 months prior to the study.
* Engaging in strenuous exercise within 48 hours prior to the tests.
* Failure to replicate the same food intake on both experimental days.
* Consumption of caffeine or any other stimulant after 6 pm on the day before the tests, to avoid headaches, discomfort, or lethargy in regular caffeine consumers.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Mean velocity at different %1RM | Through study completion, an average of 4 weeks
  Measuring bar mean velocity desplacement during bench press and back squat exercises.
Peak velocity at different %1RM | Through study completion, an average of 4 weeks
  Measuring bar peak velocity and time to reach peak velocity of bar desplacement during bench press and back squat exercises.
Mean power output at different %1RM | Through study completion, an average of 4 weeks
  Measuring during bench press and back squat exercises.
Peak power output and time to reach peak power output at different %1RM | Through study completion, an average of 4 weeks
  Measuring during bench press and back squat exercises.
Number of repetitions performed in 1 set at 65%1RM until task failure | Through study completion, an average of 4 weeks
Bar velocity deplacement performed in 1 set at 65%1RM until task failure | Through study completion, an average of 4 weeks
  In bench press and back squat exercises
Power output generated in 1 set at 65%1RM until task failure | Through study completion, an average of 4 weeks
  In bench press and back squat exercise
Muscle electrical activity (EMG). | Through study completion, an average of 4 weeks
  Root-mean-square (RMS) and maximal voluntary contraction (MVC) from pectoralis major and triceps (bench press) and from rectus femoris and vastus lateralis (Back squat).

SECONDARY OUTCOMES:
Mood state (tension, depression, anger, vigor, fatigue and confusion) | Through study completion, an average of 4 weeks
  Participants graded a set of 29 items related to the mood on a Likert scale from 0 (not at all) to 4 (extremely) in reply to the question: How do you feel at this moment? To assess six scales: tension, depression, anger, vigor, fatigue and confusion.
Adverse effects | Through study completion, an average of 4 weeks
  perception of power, endurance, energy and exertion, as well as heart, muscular and gastrointestinal discomfort.

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina y Ciencias de la Salud. Universidad de Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes